CLINICAL TRIAL: NCT06993519
Title: Effects of Minimally Non-surgical Periodontal Treatment Versus Quadrantwise Subgingival Instrumentations on Residual Periodontal Pockets
Brief Title: Impact of Minimally Non-surgical Periodontal Treatment on Residual Pockets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Gaetano Isola, Associate Professor, University of Catania
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Residual-MINST
Record Dates: First submitted 2025-05-19; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Pocket, Periodontal; Periodontitis
MeSH Terms: conditions — Periodontal Pocket; Periodontitis

STUDY DESIGN:
Intervention Model Description: Non-surgical periodontal treatment Subgingival biofilm ultrasonic debridement with MINST or Q-SI for residual pockets
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Sealed envelopes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MINST non surgical periodontal treatment (Experimental): Patients were treated with non-surgical MINST periodontal treatment in a single session on residual pockets
  Interventions: Other: Probin Pocket Depth reduction
- Q-SI non surgical periodontal treatment (Active Comparator): Periodontitis patients treated by means of Q-SI. Patients were treated with non-surgical quadrantwise periodontal treatment in 4 sessions, 1 session per week on residual pockets
  Interventions: Other: Probin Pocket Depth reduction

INTERVENTIONS:
Other: Probin Pocket Depth reduction — Probin Pocket Depth reduction in millimetres before and after treatment

SUMMARY:
A double-blind randomized-controlled clinical trial is conducted in order to evaluate the impact of non-surgical periodontal treatment by means of minimally invasive approach MINST or Q-SI (quadrantwise) approach in subjects with periodontitis on residual pockets after active periodontal treatment

DETAILED DESCRIPTION:
A double-blind randomized-controlled clinical trial is conducted in order to evaluate the impact of non-surgical periodontal treatment in subjects with periodontitis. 60 patients: 30 with periodontitis and 30 healthy controls who underwent active periodontal treatment. All the patients are assessed for clinical, periodontal, blood following of minimally invasive approach MINST or Q-SI (quadrantwise).

Measurements are taken before and after initial periodontal treatment in the periodontal subjects in order to evaluate the best treatment for residual pockets.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Periodontitis
* Presence of residula periodontal pockets

Exclusion Criteria:

* Periodontal treatment
* Use of antibiotics, NSAIDs, and immunosuppressants during the last 6 months
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-01-02 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
Probin Pocket Depth reduction | 1-year
  Probin Pocket Depth reduction in millimetres before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Isola, DDS, Principal Investigator — Università degli Studi di Catania - Dipartimento di Chirurgia Generale e Specialità Medico-Chirurgiche
Locations (1):
- Policlinico G. Rodolico, Catania, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Study results